CLINICAL TRIAL: NCT05793203
Title: Single-center Prospective Study of Non-invasive Methods for the Diagnosis of Postoperative Complications in Liver Transplant Recipients
Acronym: ElastOLT
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4176
Record Dates: First submitted 2023-03-20; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Rejection Acute Hepatic; Transplant; Failure, Liver; Liver Dysfunction
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A lot of different early and late complications may occur after liver transplantation. They could be related to surgical procedure, to infectious diseases or immuno-mediated diseases (acute cellular rejection, ACR). Almost all of those complications are characterized by an elevation in liver enzymes (ALT, AST and GGT) and a decline of liver function tests (serum bilirubin and INR increase) possibly leading to early allograft disfunction (EAD). In this scenario there is a lack of biomarker that could predict the development of ACR and/or EAD.

The aim of this study is to explore the prognostic role of non-invasive instrumental and biological marker in the early post-transplant phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for liver transplantation following National and International Guidelines

Exclusion Criteria:

* No agreement or inability to give informed consent

  * Re-transplant patients
  * Liver transplant in fulminant hepatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Allograft dysfunction (EAD) | 2 weeks from Liver transplantation
  Olthoff criteria: bilirubina≥ 10 mg/dL in 7th post-operative day, international normalized ratio (INR) ≥ 1.6 in 7th post-operative day 7; ALT or AST> 2000 IU/L during the first 7 days after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Liguori, MD, Study Chair — Catholic University of the Sacred Heart
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy